CLINICAL TRIAL: NCT02111200
Title: Comparative Efficacy of Phenylbutyrate vs. Benzoate in Urea Cycle Disorders
Brief Title: Comparative Efficacy of Phenylbutyrate (PBA) vs. Benzoate in Urea Cycle Disorders
Acronym: BPA/Benzoate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Juan Marini, Principal Investigator, Baylor College of Medicine
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: H-33157
Record Dates: First submitted 2014-04-08; First posted 2014-04-11 (Estimated); Results first posted 2017-12-08 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2017-10

CONDITIONS: Urea Cycle Disorders, Inborn
Keywords: urea cycle disorders
MeSH Terms: conditions — Urea Cycle Disorders, Inborn | interventions — Sodium Benzoate; 4-phenylbutyric acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sodium Benzoate arm (Active Comparator): Sodium benzoate 5.5 g/m2/day divided into three equal doses per day (maximum dose 12 g/day) for 3 days
  Interventions: Drug: Sodium Benzoate
- Sodium Phenylbutyrate arm (Active Comparator): Sodium phenylbutyrate 7.15 g/m2/day divided into three equal doses per day (maximum dose of 20 g/day) for 3 days
  Interventions: Drug: Sodium Phenylbutyrate
- Mix Arm (Active Comparator): Sodium Phenylbutyrate 3.575 g/m2/day and Sodium Benzoate 2.75 g/m2/day will be given in three equal doses per day for 3 days
  Interventions: Drug: Sodium Benzoate; Drug: Sodium Phenylbutyrate

INTERVENTIONS:
Drug: Sodium Benzoate — Subjects will be instructed to take the study medication with meals (08:00 breakfast; 13:00 lunch; 19:00 dinner) for 3 days.
  Arms: Mix Arm; Sodium Benzoate arm
Drug: Sodium Phenylbutyrate — Subjects will be instructed to take the study medication with meals (08:00 breakfast; 13:00 lunch; 19:00 dinner) for 3 days.
  Other Names: Buphenyl (tm)
  Arms: Mix Arm; Sodium Phenylbutyrate arm

SUMMARY:
The investigators will study and compare how effectively sodium phenylbutyrate, sodium benzoate, and a combination of the two, help excrete nitrogen in healthy volunteers. Subject participation will require three, separate, four-day study periods at least one week apart. During one study period (also called a treatment arm), subjects will take sodium phenylbutyrate; during another they will take sodium benzoate; during another they will take a combination of the two medications.

We expect to find that phenylbutyrate is more effective at removing nitrogen than benzoate or a combination of the two.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Subjects with (a) a history of frequent dietary protein intolerance, (b) a history of chronic or acute liver diseases which may result in altered hepatic synthetic capacity (e.g., hepatitis), (c) acute or chronic disease or on medications that in the opinion of the clinical investigators will interfere with the measurements (e.g., drugs which may have hepatotoxicity as potential side effects), (d) a physical disability that will interfere with their ability to either conform to the dietary regimes or undergo the isotopic infusions, (e) pregnancy or recent (<6 months)/current lactation, (f) intercurrent evidence of significant hyperammonemia (more than 100 µmol/L), (g) any clinical abnormality of Grade 3 or greater according to the Common Terminology Criteria for Adverse Events v.4.0 (CTCAE), (h) any condition(s) not covered by the CTCAE, or (i) a severe or life-threatening toxicity at screening, will be excluded from the study. Subjects taking ammonia scavenger medications will not be enrolled.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2014-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan C Marini, DVM., PhD, Principal Investigator — Baylor College of Medicine; Sandesh CS Nagamani, MD, FACMG, Principal Investigator — Baylor College of Medicine
Locations (1):
- Children's Nutrition Research Center/Baylor College of Medicine, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There was no washout period prior to enrollment. Individuals who were enrolled in the trial were not on any medications.
Groups:
- Sodium Phenylbutyrate->MIX->Sodium Benzoate (4 Days): 1. Sodium phenylbutyrate arm: Participants received ONLY sodium phenylbutyrate at a dose of 7.15 g/m2/day divided into three equal doses per day (maximum dose of 20 g/day) for 3 days. Subjects took the study medication with meals (08:00 breakfast; 13:00 lunch; 19:00 dinner) for 3 days.
     Followed by a Washout period of at least 7 days
  2. MIX arm: Participants received a combination of Sodium Phenylbutyrate 3.575 g/m2/day and Sodium Benzoate 2.75 g/m2/day were given in three equal doses per day for 3 days. Subjects took the study medications with meals (08:00 breakfast; 13:00 lunch; 19:00 dinner) for 3 days.
     Followed by a Washout period of at least 7 days
  3. Sodium benzoate: Participants received ONLY Sodium Benzoate at a dose of 5.5 g/m2/day divided into three equal doses per day (maximum dose 12 g/day) for 3 days. Subjects took the study medications with meals (08:00 breakfast; 13:00 lunch; 19:00 dinner) for 3 days.
- Sodium Benzoate->MIX-> Sodium Phenylbutyrate (4 Days): 1. Sodium benzoate: Participants received ONLY Sodium Benzoate at a dose of 5.5 g/m2/day divided into three equal doses per day (maximum dose 12 g/day) for 3 days. Subjects took the study medications with meals (08:00 breakfast; 13:00 lunch; 19:00 dinner) for 3 days.
     Followed by a Washout period of at least 7 days
  2. MIX arm: Participants received a combination of Sodium Phenylbutyrate 3.575 g/m2/day and Sodium Benzoate 2.75 g/m2/day were given in three equal doses per day for 3 days. Subjects took the study medications with meals (08:00 breakfast; 13:00 lunch; 19:00 dinner) for 3 days.
     Followed by a Washout period of at least 7 days
  3. Sodium phenylbutyrate arm: Participants received ONLY sodium phenylbutyrate at a dose of 7.15 g/m2/day divided into three equal doses per day (maximum dose of 20 g/day) for 3 days. Subjects took the study medication with meals (08:00 breakfast; 13:00 lunch; 19:00 dinner) for 3 days.
- MIX->Sodium Benzoate-> Sodium Phenylbutyrate (4 Days): 1. MIX arm: Participants received a combination of Sodium Phenylbutyrate 3.575 g/m2/day and Sodium Benzoate 2.75 g/m2/day were given in three equal doses per day for 3 days. Subjects took the study medications with meals (08:00 breakfast; 13:00 lunch; 19:00 dinner) for 3 days.
     Followed by a Washout period of at least 7 days
  2. Sodium benzoate: Participants received ONLY Sodium Benzoate at a dose of 5.5 g/m2/day divided into three equal doses per day (maximum dose 12 g/day) for 3 days. Subjects took the study medications with meals (08:00 breakfast; 13:00 lunch; 19:00 dinner) for 3 days.
     Followed by a Washout period of at least 7 days
  3. Sodium phenylbutyrate arm: Participants received ONLY sodium phenylbutyrate at a dose of 7.15 g/m2/day divided into three equal doses per day (maximum dose of 20 g/day) for 3 days. Subjects took the study medication with meals (08:00 breakfast; 13:00 lunch; 19:00 dinner) for 3 days.
- MIX-> Sodium Phenylbutyrate-> Sodium Benzoate (4 Days): 1. MIX arm: Participants received a combination of Sodium Phenylbutyrate 3.575 g/m2/day and Sodium Benzoate 2.75 g/m2/day were given in three equal doses per day for 3 days. Subjects took the study medications with meals (08:00 breakfast; 13:00 lunch; 19:00 dinner) for 3 days.
     Followed by a Washout period of at least 7 days
  2. Sodium phenylbutyrate arm: Participants received ONLY sodium phenylbutyrate at a dose of 7.15 g/m2/day divided into three equal doses per day (maximum dose of 20 g/day) for 3 days. Subjects took the study medication with meals (08:00 breakfast; 13:00 lunch; 19:00 dinner) for 3 days.
     Followed by a Washout period of at least 7 days
  3. Sodium benzoate: Participants received ONLY Sodium Benzoate at a dose of 5.5 g/m2/day divided into three equal doses per day (maximum dose 12 g/day) for 3 days. Subjects took the study medications with meals (08:00 breakfast; 13:00 lunch; 19:00 dinner) for 3 days.
Period: Overall Study
Arm/Group | Sodium Phenylbutyrate->MIX->Sodium Benzoate (4 Days) | Sodium Benzoate->MIX-> Sodium Phenylbutyrate (4 Days) | MIX->Sodium Benzoate-> Sodium Phenylbutyrate (4 Days) | MIX-> Sodium Phenylbutyrate-> Sodium Benzoate (4 Days)
Started | 3 | 2 | 1 | 1
Completed | 3 | 2 | 1 | 1
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This was a cross over design study.
Groups:
- Sodium Phenylbutyrate->MIX->Sodium Benzoate: 1. Sodium phenylbutyrate arm: Participants received ONLY sodium phenylbutyrate at a dose of 7.15 g/m2/day divided into three equal doses per day (maximum dose of 20 g/day) for 3 days. Subjects took the study medication with meals (08:00 breakfast; 13:00 lunch; 19:00 dinner) for 3 days.
     Followed by a Washout period of at least 7 days
  2. MIX arm: Participants received a combination of Sodium Phenylbutyrate 3.575 g/m2/day and Sodium Benzoate 2.75 g/m2/day were given in three equal doses per day for 3 days. Subjects took the study medications with meals (08:00 breakfast; 13:00 lunch; 19:00 dinner) for 3 days.
     Followed by a Washout period of at least 7 days
  3. Sodium benzoate: Participants received ONLY Sodium Benzoate at a dose of 5.5 g/m2/day divided into three equal doses per day (maximum dose 12 g/day) for 3 days. Subjects took the study medications with meals (08:00 breakfast; 13:00 lunch; 19:00 dinner) for 3 days.
- Sodium Benzoate->MIX-> Sodium Phenylbutyrate: 1. Sodium benzoate: Participants received ONLY Sodium Benzoate at a dose of 5.5 g/m2/day divided into three equal doses per day (maximum dose 12 g/day) for 3 days. Subjects took the study medications with meals (08:00 breakfast; 13:00 lunch; 19:00 dinner) for 3 days.
     Followed by a Washout period of at least 7 days
  2. MIX arm: Participants received a combination of Sodium Phenylbutyrate 3.575 g/m2/day and Sodium Benzoate 2.75 g/m2/day were given in three equal doses per day for 3 days. Subjects took the study medications with meals (08:00 breakfast; 13:00 lunch; 19:00 dinner) for 3 days.
     Followed by a Washout period of at least 7 days
  3. Sodium phenylbutyrate arm: Participants received ONLY sodium phenylbutyrate at a dose of 7.15 g/m2/day divided into three equal doses per day (maximum dose of 20 g/day) for 3 days. Subjects took the study medication with meals (08:00 breakfast; 13:00 lunch; 19:00 dinner) for 3 days.
- MIX->Sodium Benzoate-> Sodium Phenylbutyrate: 1. MIX arm: Participants received a combination of Sodium Phenylbutyrate 3.575 g/m2/day and Sodium Benzoate 2.75 g/m2/day were given in three equal doses per day for 3 days. Subjects took the study medications with meals (08:00 breakfast; 13:00 lunch; 19:00 dinner) for 3 days.
     Followed by a Washout period of at least 7 days
  2. Sodium benzoate: Participants received ONLY Sodium Benzoate at a dose of 5.5 g/m2/day divided into three equal doses per day (maximum dose 12 g/day) for 3 days. Subjects took the study medications with meals (08:00 breakfast; 13:00 lunch; 19:00 dinner) for 3 days.
     Followed by a Washout period of at least 7 days
  3. Sodium phenylbutyrate arm: Participants received ONLY sodium phenylbutyrate at a dose of 7.15 g/m2/day divided into three equal doses per day (maximum dose of 20 g/day) for 3 days. Subjects took the study medication with meals (08:00 breakfast; 13:00 lunch; 19:00 dinner) for 3 days.
- MIX-> Sodium Phenylbutyrate-> Sodium Benzoate: 1. MIX arm: Participants received a combination of Sodium Phenylbutyrate 3.575 g/m2/day and Sodium Benzoate 2.75 g/m2/day were given in three equal doses per day for 3 days. Subjects took the study medications with meals (08:00 breakfast; 13:00 lunch; 19:00 dinner) for 3 days.
     Followed by a Washout period of at least 7 days
  2. Sodium phenylbutyrate arm: Participants received ONLY sodium phenylbutyrate at a dose of 7.15 g/m2/day divided into three equal doses per day (maximum dose of 20 g/day) for 3 days. Subjects took the study medication with meals (08:00 breakfast; 13:00 lunch; 19:00 dinner) for 3 days.
     Followed by a Washout period of at least 7 days
  3. Sodium benzoate: Participants received ONLY Sodium Benzoate at a dose of 5.5 g/m2/day divided into three equal doses per day (maximum dose 12 g/day) for 3 days. Subjects took the study medications with meals (08:00 breakfast; 13:00 lunch; 19:00 dinner) for 3 days.
- Total: Total of all reporting groups
Arm/Group | Sodium Phenylbutyrate->MIX->Sodium Benzoate | Sodium Benzoate->MIX-> Sodium Phenylbutyrate | MIX->Sodium Benzoate-> Sodium Phenylbutyrate | MIX-> Sodium Phenylbutyrate-> Sodium Benzoate | Total
Number analyzed (Participants) | 3 | 2 | 1 | 1 | 7
Age, Continuous [Median (Full Range); unit: years] | 26 [23 to 52] | 42.5 [27 to 58] | 28 [28 to 28] | 33 [33 to 33] | 28 [23 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 1 | 2
  Male | 2 | 2 | 1 | 0 | 5
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 1 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Urinary Hippuric Acid
Description: The objective of this protocol is to directly compare the efficacy of benzoate, phenylbutyrate and a combination of the two, to conjugate nitrogenous compounds in healthy volunteers. The nitrogenous compound of interest in each arm would be based on the medication used. This would be hippuric acid in the benzoate arm, phenylacetylglutamine in the phenylbutyrate arm, and hippuric acid AND phenylacetylglutamine in the MIX arm. The mean hippuric acid levels in the phenylbutyrate arm would thus be 0.
Time Frame: 4 days per arm
Measure: Mean (Standard Deviation); unit: mmol/24 hours
Arm/Group | Sodium Benzoate Arm | Sodium Phenylbutyrate Arm | Mix Arm
Number analyzed (Participants) | 7 | 7 | 7
mmol/24 hours | 16.4 (3.1) | 0 (0) | 10.5 (1.7)

2. Primary Outcome: Urinary PAGN Excretion
Description: The objective of this protocol is to directly compare the efficacy of benzoate, phenylbutyrate and a combination of the two, to conjugate nitrogenous compounds in healthy volunteers. The nitrogenous compound of interest in each arm would be based on the medication used. This would be hippuric acid in the benzoate arm, phenylacetylglutamine in the phenylbutyrate arm, and hippuric acid AND phenylacetylglutamine in the MIX arm. The mean phenylacetylglutamine levels in the benzoate arm would thus be 0.
Time Frame: 4 days per arm
Measure: Mean (Standard Deviation); unit: mmol/24 hours
Arm/Group | Sodium Benzoate Arm | Sodium Phenylbutyrate Arm | Mix Arm
Number analyzed (Participants) | 7 | 7 | 7
mmol/24 hours | 0 (0) | 15.3 (2.3) | 9.3 (0.8)

3. Primary Outcome: Total Nitrogen as a Conjugate of the Drug
Description: The objective of this protocol is to directly compare the efficacy of benzoate, phenylbutyrate and a combination of the two, to conjugate nitrogenous compounds in healthy volunteers. The nitrogenous compound of interest in each arm would be based on the medication used. This would be hippuric acid in the benzoate arm, phenylacetylglutamine in the phenylbutyrate arm, and hippuric acid AND phenylacetylglutamine in the MIX arm.
Time Frame: 4 days per arm
Measure: Mean (Standard Deviation); unit: mmol/24 hours
Arm/Group | Sodium Benzoate Arm | Sodium Phenylbutyrate Arm | Mix Arm
Number analyzed (Participants) | 7 | 7 | 7
mmol/24 hours | 16.4 (3.1) | 29 (3.3) | 30.7 (4.5)

ADVERSE EVENTS:
Time Frame: The adverse events were collected through 4 days of each study arm.
Groups:
- Sodium Benzoate Treatment: Sodium benzoate 5.5 g/m2/day divided into three equal doses per day (maximum dose 12 g/day) for 3 days
  Sodium Benzoate: Subjects will be instructed to take the study medication with meals (08:00 breakfast; 13:00 lunch; 19:00 dinner) for 3 days.
- Sodium Phenylbutyrate Treatment: Sodium phenylbutyrate 7.15 g/m2/day divided into three equal doses per day (maximum dose of 20 g/day) for 3 days
  Sodium Phenylbutyrate: Subjects will be instructed to take the study medication with meals (08:00 breakfast; 13:00 lunch; 19:00 dinner) for 3 days.
- MIX Treatment: Sodium Phenylbutyrate 3.575 g/m2/day and Sodium Benzoate 2.75 g/m2/day will be given in three equal doses per day for 3 days
  Sodium Benzoate: Subjects will be instructed to take the study medication with meals (08:00 breakfast; 13:00 lunch; 19:00 dinner) for 3 days.
  Sodium Phenylbutyrate: Subjects will be instructed to take the study medication with meals (08:00 breakfast; 13:00 lunch; 19:00 dinner) for 3 days.
Arm/Group | Sodium Benzoate Treatment | Sodium Phenylbutyrate Treatment | MIX Treatment
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 3/7 | 5/7 | 3/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sodium Benzoate Treatment (N=7) | Sodium Phenylbutyrate Treatment (N=7) | MIX Treatment (N=7)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Lab anormalities (Investigations) | 1 (1) | 4 (8) | 2 (5)
Itch (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (General disorders) | 0 (0) | 1 (1) | 0 (0)
Toe injury (General disorders) | 1 (1) | 0 (0) | 1 (1) — Unrelated to the study procedures

LIMITATIONS AND CAVEATS:
A limitation of this study is that it was conducted in healthy subjects in whom ammonemia is well-controlled. Ammonia control was not assessed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No